CLINICAL TRIAL: NCT07323069
Title: The Dreamcatchers Programme - A Nurse-led Multicomponent Interventional Protocol to Improve Sleep Quality in Paediatric Oncology Patients: A Pilot Randomized Controlled Trial
Brief Title: A Nurse-led Multicomponent Interventional Protocol to Improve Sleep Quality in Paediatric Oncology Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Children's Hospital (Other)
Responsible Party: Principal Investigator, Mak Shuk Yan, Principal Investigator, Ward Manager (Paediatrics and Adolescent Medicine), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PAED-2025-074
Record Dates: First submitted 2025-12-03; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pediatrics Cancer
Keywords: pediatrics; oncology; leukemia; solid tumour; sleep; sleep quality; quality of life; sleep disturbances
MeSH Terms: conditions — Neoplasms; Leukemia; Sleep Initiation and Maintenance Disorders; Parasomnias | interventions — Autogenic Training; Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education with Exercises (Experimental): The intervention group will receive the Dreamcatchers Programme, including sleep hygiene education, PMR, and breathing control exercises, which will be delivered over 4 weeks with weekly in-person follow-ups.
  Interventions: Other: Sleep Hygiene Education; Other: Progressive Muscle Relaxation; Other: Breathing exercises
- Control (No Intervention): The waitlist control group will continue to receive routine hospital support and pediatric oncology health information (e.g., neutropenic diet tips) to maintain engagement without sleep-specific strategies. In order to ensure fairness, participants of the waitlist control group will be given access to the Dreamcatchers Programme once the final follow-up assessment is completed.

INTERVENTIONS:
Other: Sleep Hygiene Education — The first part of the intervention consists of a group education session on sleep hygiene. Each session will accommodate a maximum of 10 participants and will last approximately 45 minutes facilitated by a nurse using a PowerPoint presentation.
  Arms: Education with Exercises
Other: Progressive Muscle Relaxation — Following the education session, practical demonstrations of PMR will be conducted, allowing patients and caregivers to practice what they have learned. These exercises will be designed to be simple, age-appropriate, and easily integrated into daily routines.
  PMR helps lower stress and anxiety by modulating the activities of the autonomic nervous system. The entire PMR routine will take approximately 10-15 minutes, consistent with the duration of relaxation exercises noted in earlier research.
  Arms: Education with Exercises
Other: Breathing exercises — Breathing exercises will also be demonstrated and advised to be used before bedtime, aiming to reduce physiological arousal and promote relaxation through slowing down breathing rate, amplifying vagus nerve activity and normalizing stress responses. The breathing routine, incorporating box breathing techniques, will last 5-10 minutes and is to be practiced as part of the children's wind-down routine before sleep.
  Arms: Education with Exercises

SUMMARY:
Sleep is essential for a child's development, influencing cognitive function, emotional stability, recovery, and overall well-being. Prolonged and intensive treatments for pediatric oncology patients can lead to sleep disturbances that are often overlooked by caregivers and healthcare professionals as temporary side effects. Symptoms may include difficulty initiating or maintaining sleep, reduced sleep duration, or perceived poor sleep quality. Recent studies indicate that sleep disturbances affect between 13% to 50% of leukemia survivors and up to 80% of children with central nervous system tumors. A recent study in Hong Kong found that approximately 45% of pediatric oncology survivors continue to face sleep challenges, underscoring the global and local relevance of this issue.

These sleep disturbances in this vulnerable group often result from factors such as pain and nausea due to chemotherapy side effects, which can be exacerbated by corticosteroids. The immediate discomfort caused by sleep disruptions can significantly affect treatment adherence, daily activities, social interactions, and overall quality of life.

While pharmacological approaches remain the standard treatment for pediatric sleep disturbances, this method carries significant risks, including potential drug interactions and dependence. Non-pharmacological options, however, empower patients and caregivers to manage sleep issues without increasing medication use, promoting a proactive approach to sleep health.

In response to the need to enhance sleep quality among pediatric oncology patients, the Dreamcatchers Programme was developed as a nurse-led initiative. This program focuses on relaxation and offers sustainable strategies for improved sleep through sleep hygiene practices, progressive muscle relaxation (PMR), and breathing exercises for both patients and caregivers. Evidence-based interventions equip nurses with holistic techniques that address gaps in their knowledge and skills.

This project proposal details a randomized controlled pilot study aimed at evaluating the feasibility and preliminary effectiveness of the Dreamcatchers Programme, setting the groundwork for a standardized sleep management protocol in pediatric oncology care.

DETAILED DESCRIPTION:
The trial employs a prospective, single-blind, waitlist-controlled design with 1:1 allocation. Block randomization, generated by computer and concealed in sealed opaque envelopes, ensures balanced group sizes and minimizes selection and allocation bias. Blinding of participants and caregivers is infeasible due to the intervention's nature, but outcome assessors (nurses collecting data) remain blinded to group assignment to reduce observer bias.

To prevent contamination, intervention sessions occur in a separate educational room away from clinical areas. Access to supportive QR code videos of relaxation exercises is password-protected and restricted to the intervention group.

Recruitment uses simple random sampling from a computer-generated list of eligible attendees at the ambulatory chemotherapy day center of Hong Kong Children's Hospital (HKCH). Day patients are selected over inpatients for their stable attendance patterns, which support consistent intervention delivery, follow-up, and data collection. This choice enhances feasibility, aligns with the programme's intended home-based application, minimizes hospital-related confounders (e.g., interruptions, equipment), and improves generalizability to outpatient and survivorship settings.

The principal investigator approaches eligible families, obtains informed consent from caregivers, and assent from children where appropriate, reducing selection bias.

Sample size follows methodological guidance emphasizing logistical and feasibility assessments over powered hypothesis testing.

This multi-component, nurse-delivered programme targets sleep hygiene, progressive muscle relaxation (PMR), and breathing exercises.

Initial Group Education Session (~45 minutes, max 10 participants/caregivers): Nurse-facilitated PowerPoint covers sleep's role in recovery, optimal sleep environment (lighting, noise), consistent routines, screen-free alternatives, diaphragmatic breathing/PMR for relaxation, and sleep diary use (booklet for tracking habits, duration, and exercises).

Practical Demonstrations: Hands-on practice of PMR (10-15 minutes; gentle, suitable for reduced mobility/strength) and box breathing (5-10 minutes; pre-bedtime to reduce arousal via vagal stimulation).

Support Materials: QR code access to video recordings of exercises (adapted from established resources).

Weekly Follow-ups (4 weeks): Reinforcement, practice, troubleshooting, and monitoring of adherence/sleep hygiene.

Waitlist participants receive routine hospital support and general pediatric oncology education (e.g., neutropenic diet), maintaining engagement without sleep-specific content.

De-identified data (unique codes) are stored securely (password-protected files, locked physical records) per Hospital Authority policies, retained 5 years post-study, then destroyed. Incidental severe findings prompt notification while maintaining confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Children who can read and communicate in Chinese
* Aged 6 to 12 years old (school-aged children).
* Diagnosed with cancer and currently undergoing active treatment.
* Identified as experiencing sleep disturbances, defined by a Chinese Pittsburgh Sleep Quality Index (PSQI) global score of ≥5.

Exclusion Criteria:

* Diagnosed with hematological diseases unrelated to cancer (e.g., sickle cell anemia, thalassemia).
* Presence of severe cognitive impairment, which may hinder the ability to follow instructions or engage with intervention components.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality | 3 months
  The primary outcome focuses on improvements in sleep quality among pediatric oncology patients aged 6-12 years, as measured by the Chinese version of the Pittsburgh Sleep Quality Index (PSQI). PSQI score is a number from 0-21, with 0 being best and higher scores indicating worse sleep; a score over 5 suggests significant sleep problems.

SECONDARY OUTCOMES:
Overall Quality of Life | 3 months
  The secondary outcome focuses on enhancing the overall quality of life of participating children during active cancer treatment, as measured by the Chinese version of the Pediatric Quality of Life Inventory (PedsQL) Cancer Module 3.0. PedsQL score ranges from 0-100, and higher PedsQL scores indicate better quality of life.

OTHER OUTCOMES:
Acceptability | 1 month
  Additionally, the study evaluates acceptability of the programme which is assessed through a custom-designed satisfaction survey (with Likert-scale and open-ended questions) and semi-structured interviews conducted with the intervention group at T1.

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Children's Hospital, Kowloon Bay, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Some participants do not wish to share their information.

REFERENCES:
- [Background] Zupanec S, Jones H, McRae L, Papaconstantinou E, Weston J, Stremler R. A Sleep Hygiene and Relaxation Intervention for Children With Acute Lymphoblastic Leukemia: A Pilot Randomized Controlled Trial. Cancer Nurs. 2017 Nov/Dec;40(6):488-496. doi: 10.1097/NCC.0000000000000457. PMID 27922922
- [Background] Zaccaro A, Piarulli A, Laurino M, Garbella E, Menicucci D, Neri B, Gemignani A. How Breath-Control Can Change Your Life: A Systematic Review on Psycho-Physiological Correlates of Slow Breathing. Front Hum Neurosci. 2018 Sep 7;12:353. doi: 10.3389/fnhum.2018.00353. eCollection 2018. PMID 30245619
- [Background] Walter LM, Nixon GM, Davey MJ, Downie PA, Horne RS. Sleep and fatigue in pediatric oncology: A review of the literature. Sleep Med Rev. 2015 Dec;24:71-82. doi: 10.1016/j.smrv.2015.01.001. Epub 2015 Jan 13. PMID 25679070
- [Background] Teresi JA, Yu X, Stewart AL, Hays RD. Guidelines for Designing and Evaluating Feasibility Pilot Studies. Med Care. 2022 Jan 1;60(1):95-103. doi: 10.1097/MLR.0000000000001664. PMID 34812790
- [Background] Tanriverdi M, Cakir E, Akkoyunlu ME, Cakir FB. Effect of virtual reality-based exercise intervention on sleep quality in children with acute lymphoblastic leukemia and healthy siblings: A randomized controlled trial. Palliat Support Care. 2022 Aug;20(4):455-461. doi: 10.1017/S1478951522000268. PMID 35289266
- [Background] Sriasih NK, Allenidekania, Wanda D. The Effects of the COMMASH-E Intervention on the Fatigue, Sleep Quality and Functional Status of Children with Cancer in Indonesia. Compr Child Adolesc Nurs. 2019;42(sup1):197-207. doi: 10.1080/24694193.2019.1594451. PMID 31192716
- [Background] Spielman AJ, Caruso LS, Glovinsky PB. A behavioral perspective on insomnia treatment. Psychiatr Clin North Am. 1987 Dec;10(4):541-53. PMID 3332317
- [Background] Sari E, Gundogdu F, Semerci R. The Effect of Progressive Muscle Relaxation Exercises on Sleep Quality in Cancer Patients Undergoing Chemotherapy: A Randomized Controlled Study. Semin Oncol Nurs. 2024 Apr;40(2):151620. doi: 10.1016/j.soncn.2024.151620. Epub 2024 Mar 16. PMID 38494385
- [Background] Kotian PL, El-Kattan Y, Niwas S, Wu M, Lin TH, Bourdreaux B, Saini SK, Spaulding A, Kellogg-Yelder D, Parker C, Chambers-Wilson R, Bantia S, Miao Z, Williams J, Schmittou A, Raman K, Wiget PA, Chand P, Sudhakar Babu Y. Design, synthesis, and structure-activity relationships of selective biphenyl antithrombotic tissue factor/factor VIIa inhibitors. Eur J Med Chem. 2025 Sep 15;294:117708. doi: 10.1016/j.ejmech.2025.117708. Epub 2025 May 6. PMID 40378577
- [Background] Meltzer LJ, Montgomery-Downs HE, Insana SP, Walsh CM. Use of actigraphy for assessment in pediatric sleep research. Sleep Med Rev. 2012 Oct;16(5):463-75. doi: 10.1016/j.smrv.2011.10.002. Epub 2012 Mar 15. PMID 22424706
- [Background] Matricciani L, Paquet C, Galland B, Short M, Olds T. Children's sleep and health: A meta-review. Sleep Med Rev. 2019 Aug;46:136-150. doi: 10.1016/j.smrv.2019.04.011. Epub 2019 Apr 23. PMID 31121414
- [Background] Li HC, Williams PD, Williams AR, Chung JO, Chiu SY, Lopez V. Confirmatory factor analysis of the Chinese version of the Pediatric Quality-of-Life Inventory Cancer Module. Cancer Nurs. 2013 Nov-Dec;36(6):E66-72. doi: 10.1097/NCC.0b013e318276e056. PMID 23348659
- [Background] Lee S, Narendran G, Tomfohr-Madsen L, Schulte F. A systematic review of sleep in hospitalized pediatric cancer patients. Psychooncology. 2017 Aug;26(8):1059-1069. doi: 10.1002/pon.4149. Epub 2016 May 5. PMID 27147507
- [Background] da Silva Santa IN, Schveitzer MC, Dos Santos MLBM, Ghelman R, Filho VO. MUSIC INTERVENTIONS IN PEDIATRIC ONCOLOGY: Systematic review and meta-analysis. Complement Ther Med. 2021 Jun;59:102725. doi: 10.1016/j.ctim.2021.102725. Epub 2021 May 5. PMID 33964406
- [Background] Cheung YT, Brinkman TM, Mulrooney DA, Mzayek Y, Liu W, Banerjee P, Panoskaltsis-Mortari A, Srivastava D, Pui CH, Robison LL, Hudson MM, Krull KR. Impact of sleep, fatigue, and systemic inflammation on neurocognitive and behavioral outcomes in long-term survivors of childhood acute lymphoblastic leukemia. Cancer. 2017 Sep 1;123(17):3410-3419. doi: 10.1002/cncr.30742. Epub 2017 Apr 27. PMID 28452142
- [Background] Annisa, F., Allenidekania, & Chodidjah, S. (2018). Do adolescent cancer survivors need health care and psychosocial services?: An Indonesian experience. Enfermería Clínica, 28, 41-45.
- [Background] Blackwell CK, Hartstein LE, Elliott AJ, Forrest CB, Ganiban J, Hunt KJ, Camargo CA Jr, LeBourgeois MK; program collaborators for Environmental influences on Child Health Outcomes (ECHO). Better sleep, better life? How sleep quality influences children's life satisfaction. Qual Life Res. 2020 Sep;29(9):2465-2474. doi: 10.1007/s11136-020-02491-9. Epub 2020 May 12. PMID 32399666

DOCUMENTS (1):
  • Study Protocol (2025-07-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT07323069/Prot_000.pdf